CLINICAL TRIAL: NCT02861482
Title: Early Usage of Bakri Postpartum Ballon is More Effective for the Management of Postpartum Hemorrhage
Brief Title: Early Usage of Bakri Ballon in Managing Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongyu Wang (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other); Guangzhou Women and Children's Medical Center (Other); Huadu District People's Hospital of Guangzhou (Other); Shenzhen Maternity & Child Healthcare Hospital (Other); Dongguan Maternity & Child Health Hospital (Unknown); Zhuhai Maternity & Child Healthcare Hospital (Unknown); The First Maternity & Child Healthcare Hospital of Huizhou (Unknown); Nanhai Women's and Children's Hospital (Unknown); Jiangmen Maternity & Child Health Care Hospital (Unknown); The Third Affiliated Hospital of Southern Medical University (Other Government); Southern Medical University, China (Other); Zhongshan Dongsheng hospital (Unknown); Xiaolan People's Hospital of Zhongshan (Unknown); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Baoan District People's Hospital of Shenzhen (Unknown); Zengcheng District People's Hospital of Guangzhou (Unknown)
Responsible Party: Sponsor-Investigator, Dongyu Wang, M.D., First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015COOK
Record Dates: First submitted 2016-06-15; First posted 2016-08-10 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Postpartum Hemorrhage
Keywords: PPH, Bakri Ballon
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; carboprost tromethamine; Cerclage, Cervical; Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bakri Ballon (Experimental): All the enrolled patients who would undergo the laying of Bakri Balloon
  Interventions: Device: Bakri Balloon; Drug: Oxytocin; Drug: Hemabate; Drug: Duratocin; Procedure: Uterine Massage; Procedure: B-lynch Suture; Procedure: Uterine Artery Embolization using sponges; Procedure: Cervical cerclage; Procedure: Hysterectomy; Drug: Blood Product

INTERVENTIONS:
Device: Bakri Balloon — Gradually increase the liquid volume inside Bakri Balloon to 250-500ml until bleeding is decreased or stopped
Drug: Oxytocin — using oxytocin(usage:20IU oxytocin in 500ml lactated Ringer's, ivgtt to a maximum of 60IU) for the first step when dealing with PPH before laying Bakri Balloon
Drug: Hemabate — using Hemabate (usage:250-500ug im) for the first step when dealing with PPH before laying Bakri Balloon
Drug: Duratocin — using Duratocin (usage:100ug iv) for the first step when dealing with PPH before laying Bakri Balloon
Procedure: Uterine Massage — continuous uterine massage for the first step when dealing with PPH before laying Bakri Balloon
Procedure: B-lynch Suture — One of conservative surgical procedures if Bakri Balloon didn't work
Procedure: Uterine Artery Embolization using sponges — One of conservative surgical procedures if Bakri Balloon didn't work
Procedure: Cervical cerclage — One of conservative surgical procedures if Bakri Balloon didn't work
Procedure: Hysterectomy — Hysterectomy with all the above measures not working
Drug: Blood Product — transfusion of blood product if necessary no matter which surgical procedure has been taken

SUMMARY:
Postpartum hemorrhage (PPH) is the top reason for maternal deaths in China. The four major causes of PPH include uterine atony, genital tract laceration, placenta factors and systemic medical disorders (including inherited and acquired coagulopathy). Management of PPH contains the application of uterotonic agents, using hemostasis agents, transfusion of blood component products, conservative procedures (intrauterine packing or balloon tamponade, compression sutures, vascular ligation and uterine artery embolization using sponges), and even hysterectomy.

The Bakri Balloon has attained its efficacy and popularity ever since it was invented by Doctor YN. Bakri. Although it is recommended by many countries as a routine procedure for PPH management, the Bakri Balloon is not yet a first choice in China due to lack in clinical data of preventive usage.

The aim of this study is to prove the efficacy and safety of the Bakri Balloon in early management of PPH.

DETAILED DESCRIPTION:
Data of 472 patients from 20 different hospitals had a Bakri balloon tamponade. Enrolled patients would follow the next process: assessment of blood loss intrapartum and 2 hours postpartum; laying the Bakri Balloon; assessment of blood loss, uterine contraction and complications after Bakri Balloon tamponade; further conservative surgical measures (uterine placation (B-lynch suture), arterial embolization; artery ligation; cervical cerclage) or even hysterectomy if necessary; recording the puerperium infection and involution of uterus.

Data were analyzed by SPSS 20.0 database. The results were expressed as mean ± standard deviations or median with interquartile range. Differences between groups were assessed by Student's unpaired t test, Mann-Whitney U test, or Chi-square test as appropriate. Correlation analysis was performed using the Spearman rank correlation method. To identify independent relationships and adjust the effects of covariates, multiple linear regression analyses were performed. P values of <0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Women with vaginal or cesarean delivery;
* PPH caused by: Uterine Atony, Placenta Factors, Coagulation disorders, Hematological disorders, Hepatic diseases, Obstetric DIC;
* Not reacting well to continuous uterine massage or uterotonic agents including oxytocin (0.04IU/L ivgtt to a maximum of 60IU), Hemabate (250-500ug im) and Duratocin (100ug iv);

  * Without other conservative surgical treatment(uterine compression suture, internal arterial embolism; vascular ligation);
* Signing the informed consents;

Exclusion Criteria:

* Has undergone or will undergo conservative surgical treatment(uterine compression suture, international arterial embolism; artery ligation);
* Impaired soft birth canal injury;
* Untreated uterine deformity;
* Definite indication for uterectomy.

Ages: 19 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 472 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Blood loss after Bakri Ballon temponade | from using Bakri Ballon Temponade to remove of Bakri Balloon Temponade with the interval ranging from 24hrs to 51hrs

SECONDARY OUTCOMES:
Ratio of Bakri Ballon only without other invasive measures in succeeding controlling PPH to the number of cases | From delivery to remove of Bakri Balloon Temponade with the interval ranging from 24hrs to 51hrs

CONTACTS AND LOCATIONS:
Overall Officials: Zilian Wang, M.D.,PhD, Study Director — Obstetrics and Gynechology Department of the 1st affiliated hospital of Sun Yat-sen University
Locations (1):
- Obstetrics and Gynechology Department of the 1st affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No